CLINICAL TRIAL: NCT07348640
Title: A Prospective, Multi-National, Randomized, Double-Blind, Crossover Study to Evaluate the Efficacy and Safety of Gadopiclenol-enhanced MRA Compared to Gadoterate Meglumine-enhanced MRA in the Assessment of Steno-occlusive Disease in Adult Patients With Suspected Vascular Disease
Brief Title: Evaluation of the Efficacy and Safety of Magnetic Resonance Angiography (MRA) Using Gadopiclenol Compared to Gadoterate Meglumine in the Assessment of Steno-occlusive Disease in Adult Patients With Suspected Vascular Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guerbet (Industry)
Collaborators: Bracco Imaging S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: GDX-102 - GDX-44-017; 2024-518835-13-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Steno-occlusive Disease
Keywords: steno-occlusive disease; gadopiclenol; Magnetic Resonnance Angiography
MeSH Terms: interventions — gadopiclenol; gadoterate meglumine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AB (Experimental): Gadopiclenol administered first followed by Gadoterate meglumine 0.1 mmol/kg
  Interventions: Drug: gadopiclenol; Drug: Gadoterate meglumine (Dotarem)
- BA (Active Comparator): Gadoterate meglumine 0.1 mmol/kg administered first followed by Gadopiclenol
  Interventions: Drug: gadopiclenol; Drug: Gadoterate meglumine (Dotarem)

INTERVENTIONS:
Drug: gadopiclenol — Gadopiclenol enhanced-Magnetic Resonance Angiography
Drug: Gadoterate meglumine (Dotarem) — Gadoterate meglumine (Dotarem) enhanced-Magnetic Resonance Angiography

SUMMARY:
Compare the diagnostic performance of gadopiclenol against gadoterate meglumine in patients with vascular diseases of supra-aortic, peripheral, or abdominal / renal arteries using MRI

DETAILED DESCRIPTION:
To prospectively compare the diagnostic performance of gadopiclenol with gadoterate meglumine given at a dose of 0.1 mmol/kg in the diagnosis and evaluation of vascular diseases of supra-aortic (carotid/vertebrobasilar), peripheral or abdominal/renal arteries using commercial MRI scanners and MRA sequences.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years of age or older willing to participate in the trial and follow all study procedures specified in the protocol.
2. Patient having read the information in the ICF and having provided his/her consent to participate in writing by dating and signing the ICF prior to any trial related procedure being conducted.
3. Patient with suspected steno-occlusive disease in supra-aortic (carotid/vertebrobasilar) (a), peripheral (b) or abdominal/renal (c) arteries based on:

   1. clinical signs and symptoms including but not limited to prior stroke, transient ischemic attack (TIA), amaurosis fugax (transient monocular blindness) and/or previous diagnostic tests (CTA, IA-DSA, or ultrasound) or
   2. symptoms of lower-extremity arterial disease (stages II-IV according to the Leriche-Fontaine classification, or 1 to 6 according to Rutherford classification 113 and/or confirmed by previous imaging (Doppler ultrasound, CTA, MRA, IADSA) or
   3. suspected renovascular hypertension based on one or more of the following criteria:

   i. hypertension refractory to standard therapy ii. acute worsening of pre-existing hypertension iii. abrupt onset of sustained, moderate to severe hypertension at age <35 years suggestive of fibromuscular dysplasia (FMD) iv. progressive renal insufficiency (creatinine > 2 mg/dL; no other apparent cause of progressive renal failure based on routine medical history, physical examination, 24-h urine collection and urinary protein excretion) v. abnormal/inconclusive renal doppler ultrasound. vi. other criteria (to be specified)
4. Are scheduled for or had undergone CTA and/or IA-DSA according to imaging standards to cover the supra-aortic (carotid/vertebrobasilar) and/or peripheral and/or abdominal/renal territory described in this protocol.

Exclusion Criteria:

1. Is a pregnant or lactating female. Exclude the possibility of pregnancy for women of childbearing potential:

   * by testing on site at the institution (serum βHCG or urine)
   * by surgical history (e.g., tubal ligation or hysterectomy)
   * post-menopausal with a minimum 1 year without menses.
2. Has any known allergy to one or more of the ingredients in the investigational products or has a history of hypersensitivity to other GBCAs.
3. Has severe renal impairment defined as an estimated glomerular filtration rate (eGFR) below 30 mL/min/1.73 m2 calculated using the Modification of Diet in Renal Disease (MDRD) formula.
4. Has known or suspected acute kidney injury (AKI) based on: a. Increase in serum creatinine by ≥ 0.3 mg/dL (≥ 26.5 μmol/L) within 48 hours or b. Increase in serum creatinine to ≥ 1.5 times baseline, which is known or presumed to have occurred within prior 7 days or c. Urine volume < 0.5 mL/kg/h for 6 hours
5. Has received any contrast agent (for MRI, CT, DSA) prior to the first IMP administration or is scheduled to receive any contrast agent between the two MRA or after the second IMP administration.
6. Has received or is scheduled for therapeutic intervention (e.g., endovascular therapy, vascular surgery, etc.) of any kind for vascular disease in the arterial territory of interest performed between the 2 MRA procedures or between the study MRAs and the CTA/IADSA procedures when applicable.
7. Has any contraindications to MRI.
8. Is suffering from severe claustrophobia.
9. Has received an investigational drug or medical device before admission into this study or scheduled to receive any investigational treatment in the course of the trial.
10. Was previously included in this trial.
11. Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority | 30 days
  To demonstrate the non-inferiority of gadopiclenol-enhanced Magnetic Resonance Angiography (MRA) compared to gadoterate meglumine enhanced MRA at 0.1 mmol/kg body weight in terms of sensitivity and specificity for detecting clinically significant steno-occlusive disease at segment level using Computerized Tomography Angiography (CTA) and/or Intra-arterial-Digital Subtraction Angiography (IA-DSA) findings as Standard of Truth.

SECONDARY OUTCOMES:
Adverse Events | 30 days
  To assess the safety profile of gadopiclenol and gadoterate meglumine 0.1 mmol/kg in terms of incidence of adverse events and changes in vital signs.

CONTACTS AND LOCATIONS:
Locations (41):
- United States (6):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Northshore - Evanston Hospital, Evanston, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Houston Methodist Hospital, Houston, Texas
  - University of Washington, Seattle, Washington
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada
- Czechia (2):
  - Department of Radiology and Nuclear Medicine, University Hospital Brno, Brno
  - Motol University Hospital, Prague
- France (4):
  - CHU Hopitaux de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital Cardiovasculaire et Pneumologique, Bron
  - CHU Dijon Bourgogne, Dijon
  - CHU de Poitiers, Poitiers
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - University Hospital Bonn, Bonn
  - UH Essen, Essen
  - University Hospital of Saarland, Homburg
  - Klinik fuer Diagnostische Radiologie and Neuroradiologie, Kiel
  - Department of Neuroradiology, UKSH Campus Lübeck, Lübeck
  - LMU University Hospital, München
- Hungary (3):
  - Semmelweis University - Budapest, Budapest
  - University of Debrecen - Debrecen, Debrecen
  - University of Pecs Clinical Centre, Pécs
- Italy (7):
  - Reparto di Neuroradiologia ASST Ospedale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera di Monserrato, Cagliari
  - ITAB -Institute of Advanced Biomedical Technologies University d'Annunzio of Chieti-Pescara, Chieti
  - Department of Diagnostic Imaging, Humanitas Research Hospital, Milan
  - Diagnostica per Immagini e Interventistica Ospedale Umberto I, Roma
  - Catholic University - Fondazione Policlinico Gemelli Advanced Radiology Center - Diagnostic Imaging and Oncologic Radiotherapy Dept. IRCCS Rome, Roma
  - Ospedale Ca' Foncello, Treviso
- Poland (3):
  - University Hospital No.1, Department of Radiology and Diagnostic Imagine, Bydgoszcz
  - Radiology Department, Uniwersyteckie Centrum Kliniczne w Gdansku, Gdansk
  - Medical University Lublin, Diagnostic Imaging Department, Lublin
- South Korea (5):
  - Yonsei University Gangnam Severance Hospital, Seoul, Gangnam-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Seoul St. Mary's Hospital, Seoul, Seocho-gu
  - Asan Medical Center, Seoul, Songpa-gu
  - Ajou University Hospital, Gyeonggi-do, Suwon-si
- Spain (3):
  - Diagnòstic per la Imatge, Barcelona
  - Hospital Clínico San Cecilio, Granada
  - Hospital Nuestra, Resonancia Magnetica NTRA, Madrid

IPD SHARING:
Plan to Share IPD: No